CLINICAL TRIAL: NCT04981379
Title: Efficacy and Safety of the Use of Hydroxychloroquine, Favipiravir or Hydroxychloroquine + Favipiravir in Early SARS-CoV-2 (COVID-19) Treatment
Brief Title: Clinical Trial For Early SARS-CoV-2 (COVID-19) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Health Institutes of Turkey (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COVID-19-FAV-HQ
Record Dates: First submitted 2021-07-26; First posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-06

CONDITIONS: Covid19
Keywords: COVID-19; Hydroxychloroquine; Favipiravir
MeSH Terms: conditions — COVID-19 | interventions — Hydroxychloroquine; favipiravir

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hydroxychloroquine + Favipiravir (Active Comparator): Hydroxychloroquine 2x200 mg 5 days and favipiravir 2 x 1600 mg loading, then 4 days 2 x 600 mg maintenance (5 days)
  Interventions: Drug: Favipiravir + Hydroxychloroquine
- Favipiravir + Placebo (Hydroxychloroquine) (Active Comparator): Favipiravir 2 x 1600 mg loading, then 4 days 2 x 600 mg maintenance (5 days) + Placebo (Hydroxychloroquine ) 2x200 mg (5 days)
  Interventions: Drug: Favipiravir
- Hydroxychloroquine + Placebo (Favipiravir) (Active Comparator): Hydroxychloroquine 2x200 mg (for 5 days) + placebo (favipiravir) 2 x 1600 mg loading, then 4 days 2 x 600 mg maintenance (5 days)
  Interventions: Drug: Hydroxychloroquine
- Placebo (Favipiravir) + Placebo (Hydroxychloroquine) (Placebo Comparator): Placebo (favipiravir) 2 x 1600 mg loading, then 4 days 2 x 600 mg maintenance (5 days) + Placebo (Hydroxychloroquine) 2x200 mg (5 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine (200 mg), as two tablets per day for 5-day interval + Placebo [Favipiravir (1600 mg)], as two tablet per day at the first day and then Favipiravir (600 mg) as two tablet per day for the remaining 4-day interval.
  Other Names: Hydroxychloroquine sulfate
  Arms: Hydroxychloroquine + Placebo (Favipiravir)
Drug: Favipiravir — Favipiravir (1600 mg), as two tablet per day at the first day and then Favipiravir (600 mg) as two tablet per day for the remaining 4-day interval + Placebo [Hydroxychloroquine (200 mg)], as two tablets per day for 5-day interval.
  Other Names: Favicovir Film Tablet
  Arms: Favipiravir + Placebo (Hydroxychloroquine)
Drug: Favipiravir + Hydroxychloroquine — Favipiravir (1600 mg), as two tablet per day at the first day and then Favipiravir (600 mg) as two tablet per day for the remaining 4-day interval + Hydroxychloroquine (200 mg), as two tablets per day for 5-day interval.
  Other Names: Favicovir Film Tablet + Hydroxychloroquine sulfate
  Arms: Hydroxychloroquine + Favipiravir
Drug: Placebo — Placebo [Favipiravir (1600 mg)], as two tablet per day at the first day and then Placebo Favipiravir (600 mg) as two tablet per day for the remaining 4-day interval + Hydroxychloroquine (200 mg), as two tablets per day for 5-day interval.
  Arms: Placebo (Favipiravir) + Placebo (Hydroxychloroquine)

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase III clinical trial which aims to investigate the superiority of hydroxychloroquine, favipiravir or hydroxychloroquine + favipiravir treatment, initiated especially in the early period in the treatment of COVID-19, over the patients being followed up with placebo in adults aged 18~59 Years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, and placebo controlled phase III clinical trial in in adults aged 18~59 Years. The study was planned as a multicenter, randomized controlled, double-blind, parallel-arm drug study. The purpose of this study is to evaluate the efficacy and safety of hydroxychloroquine, favipiravir, or hydroxychloroquine + favipiravir treatments that were initiated early in patients who were caught during filiation or who were decided to be outpatient due to mild disease findings during hospital admission, after the diagnosis of COVID-19 against patients with placebo. It is planned that the study will be conducted with two separate arms. Study arms are planned as 2:2:2:1 for 320:320:320:160 patients as follows. The dose of Favipiravir has been determined as the standard dose. Hydroxychloroquine will also be given without a loading dose.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who have understood all the procedures to be applied within the scope of the study protocol and gave their consent.
2. Patients between 18-60 years old.
3. Patients whose symptoms and complaints associated with COVID-19 started within 48 hours.
4. Mild cases whose treatment to be given as outpatient.

   1. Although asymptomatic, patients with high CRP (> 20 mg/L) and/or lymphopenia (<1000/mm3)
   2. Patients with symptoms such as fever, muscle/joint pain, cough, sore throat, nasal congestion, loss of smell.
   3. Patients without serious underlying diseases (cardiovascular diseases, diabetes mellitus, hypertension, cancer, chronic lung diseases, immunosuppressive conditions)
   4. Patients with normal chest x-ray and / or chest tomography (no sign of pneumonia)
5. Patients who accept oropharyngeal sample and venous blood collection at regular intervals within the scope of the protocol.
6. Patients who were not involved in any other interventional study.

Exclusion Criteria:

1. Patients who do not give their consent in writing after informing.
2. Being under the age of 18 and over the age of 60.
3. Patients with a known history of allergy to one of the study drugs (hydroxychloroquine, favipiravir).
4. Volunteers who the researcher thinks may have problems with adherence to treatment.
5. Volunteers who will have trouble taking medication by mouth due to resistant nausea, vomiting or chronic diarrhea.
6. Patients with chronic liver disease and transaminase (ALT or AST) levels 5 times the higher than the normal level.
7. Patients with heart disease or arrhythmia history.
8. Patients with gout or hyperuricemia.
9. Patients with signs of pneumonia in their lungs.
10. Patients with chronic renal failure (glomerular filtration rate <30).
11. Pregnant or breastfeeding patients.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1120 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-16 (Actual)

PRIMARY OUTCOMES:
Worsening of clinical findings | During the study
  Worsening of clinical findings such as respiratory distress or persistence of fever, which require hospital admission to begin another treatment (for example, remdesivir, dexamethasone, anti-cytokines, etc.)

SECONDARY OUTCOMES:
Complete resolution of symptoms and signs | Fifth day after examination
  Complete resolution of symptoms and signs
Complete resolution of symptoms and signs | Tenth day after examination
  Complete resolution of symptoms and signs
Negative RT-PCR test for SARS-CoV-2 | Tenth day after examination
  Negative RT-PCR test for SARS-CoV-2 virus
Determination of IgM, IgG levels for SARS-CoV-2 | Tenth day after examination
  Determination of IgM, IgG levels for SARS-CoV-2 virus
Negative RT-PCR test for SARS-CoV-2 | Thirtieth day after examination
  Negative RT-PCR test for SARS-CoV-2 on the 30th day visit
Determination of IgM, IgG antibodies | Thirtieth day after examination
  Determination of IgM, IgG antibodies against SARS-CoV-2
Development of signs of pneumonia | During the study
  Development of signs of pneumonia
Requirement of respiratory support with oxygen mask | During the study
  Requirement of respiratory support with oxygen mask
Requirement of respiratory support with high flow oxygen | During the study
  Requirement of respiratory support with high flow oxygen
Requirement of mechanical ventilation | During the study
  Requirement of mechanical ventilation
Death | During the study
  Death
The rate of discontinuation of treatments due to side effects | During the study
  The rate of discontinuation of treatments due to side effects (gastrointestinal, allergic skin rash, arrhythmia, other cardiac reasons)
Time to improvement of symptoms after the initiation of study drugs | During the study
  Time to improvement of symptoms after the initiation of study drugs

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Gül, Prof., Study Director — Faculty Member
Locations (6):
- Turkey (Türkiye) (6):
  - Ankara City Hospital, Ankara
  - Başakşehir Çam ve Sakura City Hospital, Istanbul
  - Istanbul Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul
  - Istanbul University Istanbul Medicine Faculty, Istanbul
  - Kartal Dr. Lütfi Kırdar City Hospital, Istanbul
  - Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCullough PA. Favipiravir and the Need for Early Ambulatory Treatment of SARS-CoV-2 Infection (COVID-19). Antimicrob Agents Chemother. 2020 Nov 17;64(12):e02017-20. doi: 10.1128/AAC.02017-20. Print 2020 Nov 17. PMID 32967849
- [Background] Shrestha DB, Budhathoki P, Khadka S, Shah PB, Pokharel N, Rashmi P. Favipiravir versus other antiviral or standard of care for COVID-19 treatment: a rapid systematic review and meta-analysis. Virol J. 2020 Sep 24;17(1):141. doi: 10.1186/s12985-020-01412-z. PMID 32972430
- [Background] Doi Y, Hibino M, Hase R, Yamamoto M, Kasamatsu Y, Hirose M, Mutoh Y, Homma Y, Terada M, Ogawa T, Kashizaki F, Yokoyama T, Koba H, Kasahara H, Yokota K, Kato H, Yoshida J, Kita T, Kato Y, Kamio T, Kodama N, Uchida Y, Ikeda N, Shinoda M, Nakagawa A, Nakatsumi H, Horiguchi T, Iwata M, Matsuyama A, Banno S, Koseki T, Teramachi M, Miyata M, Tajima S, Maeki T, Nakayama E, Taniguchi S, Lim CK, Saijo M, Imai T, Yoshida H, Kabata D, Shintani A, Yuzawa Y, Kondo M. A Prospective, Randomized, Open-Label Trial of Early versus Late Favipiravir Therapy in Hospitalized Patients with COVID-19. Antimicrob Agents Chemother. 2020 Nov 17;64(12):e01897-20. doi: 10.1128/AAC.01897-20. Print 2020 Nov 17. PMID 32958718
- [Background] Hu TY, Frieman M, Wolfram J. Insights from nanomedicine into chloroquine efficacy against COVID-19. Nat Nanotechnol. 2020 Apr;15(4):247-249. doi: 10.1038/s41565-020-0674-9. PMID 32203437
- [Background] Boulware DR, Pullen MF, Bangdiwala AS, Pastick KA, Lofgren SM, Okafor EC, Skipper CP, Nascene AA, Nicol MR, Abassi M, Engen NW, Cheng MP, LaBar D, Lother SA, MacKenzie LJ, Drobot G, Marten N, Zarychanski R, Kelly LE, Schwartz IS, McDonald EG, Rajasingham R, Lee TC, Hullsiek KH. A Randomized Trial of Hydroxychloroquine as Postexposure Prophylaxis for Covid-19. N Engl J Med. 2020 Aug 6;383(6):517-525. doi: 10.1056/NEJMoa2016638. Epub 2020 Jun 3. PMID 32492293
- [Background] Kaptein SJF, Jacobs S, Langendries L, Seldeslachts L, Ter Horst S, Liesenborghs L, Hens B, Vergote V, Heylen E, Barthelemy K, Maas E, De Keyzer C, Bervoets L, Rymenants J, Van Buyten T, Zhang X, Abdelnabi R, Pang J, Williams R, Thibaut HJ, Dallmeier K, Boudewijns R, Wouters J, Augustijns P, Verougstraete N, Cawthorne C, Breuer J, Solas C, Weynand B, Annaert P, Spriet I, Vande Velde G, Neyts J, Rocha-Pereira J, Delang L. Favipiravir at high doses has potent antiviral activity in SARS-CoV-2-infected hamsters, whereas hydroxychloroquine lacks activity. Proc Natl Acad Sci U S A. 2020 Oct 27;117(43):26955-26965. doi: 10.1073/pnas.2014441117. Epub 2020 Oct 9. PMID 33037151